CLINICAL TRIAL: NCT03085017
Title: Effectiveness of BoneSeal® on Bone Hemostats in Patients Undergoing Cardiothoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5160386; 16042 (Other: Loma Linda Clinial Trials Center)
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Results first posted 2020-09-22 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Bypass Grafting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ostene (Active Comparator): Application of Ostene onto cut sternal site for hemostasis.
  Interventions: Device: Ostene
- BoneSeal (Experimental): Application of BoneSeal onto cut sternal site for hemostasis.
  Interventions: Device: BoneSeal

INTERVENTIONS:
Device: BoneSeal — BoneSeal® is an absorbable synthetic bone hemostats that also contains of PLA, PEG and hydroxyapatite which supports bone re-growth. Product code MTJ. FDA number K142348.
  Arms: BoneSeal
Device: Ostene — OSTENE is a synthetic, biodissolvable implant material that, provides immediate bone hemostasis, can be used on all bleeding bone surfaces, is completely biocompatible and water-soluble polymer, is a mechanical barrier that does not act biochemically.
  Arms: Ostene

SUMMARY:
A prospective randomized open-label study that will evaluate the effectiveness of the pliable and absorbable bone hemostats (BoneSeal®) on the reduction of bleeding from the sternal bone marrow in patients undergoing cardiothoracic surgery.

DETAILED DESCRIPTION:
A prospective randomized open-label study that will evaluate the effectiveness of the pliable and absorbable bone hemostats (BoneSeal®) composed of synthetic materials and hydroxyapatite on the reduction of bleeding from the sternal bone marrow in patients undergoing Coronary Artery Bypass Grafting, with or without valve replacement or repair. This product will be compared to the similar, currently used product, Ostene®. Bleeding will be evaluated qualitatively by the surgeon as well as quantitatively by comparing pre- and post-operative hemoglobin levels, intra-operative and post-operative blood product usage, and post-operative chest tube output. A 30 day follow-up will be conducted to evaluate the patient's tolerance of the product, possible complications, or infection. Additionally, surgeons will be asked to comment on the ease of use of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Consent given by patient prior to surgery
2. Adult patients over 45 years
3. Subjects requiring elective, prescheduled or urgent open heart surgery requiring a sternotomy including, but not limited to CABG, valve repair, valve replacement

Exclusion Criteria:

1. An immune system disorder
2. Known hypersensitivity to components in BoneSeal® or Ostene®
3. Patients undergoing emergency surgery
4. Patients undergoing aortic dissection
5. No consent given

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Rabkin, MD, FACS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Light R. Hemostasis in neurosurgery. Journal of neurosurgery. 1945; 2(5): p. 414-34.
- [Background] Nelson DR, Buxton TB, Luu QN, Rissing JP. The promotional effect of bone wax on experimental Staphylococcus aureus osteomyelitis. J Thorac Cardiovasc Surg. 1990 Jun;99(6):977-80. PMID 2359338
- [Background] Sudmann B, Bang G, Sudmann E. Histologically verified bone wax (beeswax) granuloma after median sternotomy in 17 of 18 autopsy cases. Pathology. 2006 Apr;38(2):138-41. doi: 10.1080/00313020600561732. PMID 16581654
- [Background] Johnson P, Fromm D. Effects of bone wax on bacterial clearance. Surgery. 1981 Feb;89(2):206-9. PMID 7006134
- [Background] Orgill DP, Ehret FW, Regan JF, Glowacki J, Mulliken JB. Polyethylene glycol/microfibrillar collagen composite as a new resorbable hemostatic bone wax. J Biomed Mater Res. 1998 Mar 5;39(3):358-63. doi: 10.1002/(sici)1097-4636(19980305)39:33.0.co;2-i. PMID 9468043
- [Background] Solheim E, Pinholt EM, Andersen R, Bang G, Sudmann E. The effect of a composite of polyorthoester and demineralized bone on the healing of large segmental defects of the radius in rats. J Bone Joint Surg Am. 1992 Dec;74(10):1456-63. PMID 1469005
- [Background] Solheim E, Pinholt EM, Bang G, Sudmann E. Effect of local hemostatics on bone induction in rats: a comparative study of bone wax, fibrin-collagen paste, and bioerodible polyorthoester with and without gentamicin. J Biomed Mater Res. 1992 Jun;26(6):791-800. doi: 10.1002/jbm.820260608. PMID 1527101
- [Background] Sugamori T, Iwase H, Maeda M, Inoue Y, Kurosawa H. Local hemostatic effects of microcrystalline partially deacetylated chitin hydrochloride. J Biomed Mater Res. 2000 Feb;49(2):225-32. doi: 10.1002/(sici)1097-4636(200002)49:23.0.co;2-v. PMID 10571909
- [Background] Wilkinson HA, Baker S, Rosenfeld S. Gelfoam paste in experimental laminectomy and cranial trephination: hemostasis and bone healing. J Neurosurg. 1981 May;54(5):664-7. doi: 10.3171/jns.1981.54.5.0664. PMID 7229706
- [Background] Magyar CE, Aghaloo TL, Atti E, Tetradis S. Ostene, a new alkylene oxide copolymer bone hemostatic material, does not inhibit bone healing. Neurosurgery. 2008 Oct;63(4 Suppl 2):373-8; discussion 378. doi: 10.1227/01.NEU.0000316859.03788.44. PMID 18981846
- [Background] Vestergaard RF, Bruel A, Thomsen JS, Hauge EM, Soballe K, Hasenkam JM. The influence of hemostatic agents on bone healing after sternotomy in a porcine model. Ann Thorac Surg. 2015 Mar;99(3):1005-11. doi: 10.1016/j.athoracsur.2014.10.016. Epub 2015 Jan 16. PMID 25601654
- [Background] Higashi S, Yamamuro T, Nakamura T, Ikada Y, Hyon SH, Jamshidi K. Polymer-hydroxyapatite composites for biodegradable bone fillers. Biomaterials. 1986 May;7(3):183-7. doi: 10.1016/0142-9612(86)90099-2. PMID 3013326
- [Background] Overgaard S, Soballe K, Lind M, Bunger C. Resorption of hydroxyapatite and fluorapatite coatings in man. An experimental study in trabecular bone. J Bone Joint Surg Br. 1997 Jul;79(4):654-9. doi: 10.1302/0301-620x.79b4.7670. PMID 9250760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ostene | BoneSeal
Started | 30 | 27
Completed | 30 | 24
Not Completed | 0 | 3
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: 30 subjects had Ostene applied on cut sternal bone site. 27 subjects had BoneSeal applied on cut sternal bone site.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ostene | BoneSeal | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.7) | 60.0 (8.0) | 64.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 1 | 1 | 2
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use
Description: Qualitative determination of product application and hemostatic qualities graded by the surgeon using a scale from 1-5 with 1 being very easy and 5 being very difficult
Time Frame: The time frame for assessing the ease of product application is the short interval a the conclusion of the operation when we are applying the topical hemostatic agent to the sternal bone marrow. In other words at the end of the case, this takes <10 min.
Population: Subjects undergoing Coronary Artery Bypass Grafting with or without valve replacement repair requiring hemostatic product for cut sternal bone site.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
units on a scale | 4 [1 to 5] | 1 [1 to 3]

2. Primary Outcome: Number of Participants Experiencing Re-bleed
Description: Occurrence of re-bleeding during the operation will be noted. Reapplication of product will not occur.
Time Frame: 0-3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
Participants | 25 | 3

3. Primary Outcome: Hemoglobin
Description: Postoperative hemoglobin as compared to baseline preoperative readings
Time Frame: Pre-operative (baseline) and Post-operative (3-6 hours after baseline)
Population: Subjects undergoing Coronary Artery Bypass Grafting, with or without valve replacement or repair and needing hemostatic products be used on cut sternal bone site.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
g/dL
  Pre-operative Hemoglobin | 12.7 (2.1) | 12.7 (2.1)
  Post-operative hemoglobin | 9.9 (2.0) | 10.9 (2.1)

4. Primary Outcome: Intra-operative Blood Units
Description: Units of blood/blood products transfused during surgery
Time Frame: 0-3 hours
Measure: Mean (Standard Deviation); unit: Blood Units
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
Blood Units | 0.50 (0.96) | 0.26 (.81)

5. Primary Outcome: Surgical Site Drainage
Description: Post-operative chest tube output
Time Frame: 6, 12, 18 and 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
mL
  6 Hour | 309.3 (245.1) | 294.3 (245.1)
  12 Hour | 463.7 (338.7) | 439.3 (338.7)
  18 Hour | 598.4 (380.6) | 568.3 (380.6)
  24 Hour | 683.5 (409.5) | 647.1 (409.5)

6. Primary Outcome: Number of Participants With Post Operative Complications Related to the Device
Description: Sternal wound infection or other complications related to the device or its use within 30 days post procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 24
Participants | 2 | 0

7. Primary Outcome: Number of Participants Requiring Use of Another Product During Surgery
Description: The surgeon's determination and need for the use of another product (FloSeal) during surgery to stop bleeding or re-bleed at the sternum.
Time Frame: During surgery, up to 3 hours
Population: Subjects undergoing Coronary Artery Bypass Grafting, with or without valve replacement or repair and in need of a hemostatic agent be applied on cut sternal bone site.
Measure: Count of Participants; unit: Participants
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
Participants | 13 | 1

8. Primary Outcome: End of Surgery Bleeding
Description: Qualitative determination of of the amount of bleeding at the sternum at the end of surgery by the surgeon using a scale from 1-5 with 1 none and 5 being perfuse
Time Frame: End of surgery (closure of the chest)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
units on a scale | 4 [1 to 5] | 2 [1 to 3]

9. Primary Outcome: Post-operative Blood Units
Description: Units of blood/blood products transfused within 24 hours post surgery
Time Frame: 3-24 hours
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Blood Units
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 27
Blood Units | 0.50 (0.96) | 0.26 (0.81)

10. Primary Outcome: Number of Participants With Infection
Description: The presence of an infection at the sternum at any time up to 30 days post surgery.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ostene | BoneSeal
Number analyzed (Participants) | 30 | 24
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Ostene | BoneSeal
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/27
Other Adverse Events (participants affected / at risk) | 1/30 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ostene (N=30) | BoneSeal (N=27)
Infection (Surgical and medical procedures) | 1 (1) | 0 (0) — Deep sternal wound infection. There were no adverse events in the BoneSeal group.
OTHER ADVERSE EVENTS (reported when occurring in more than 3.33% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ostene (N=30) | BoneSeal (N=27)
keloid formation at sternum (Surgical and medical procedures) | 1 (1) | 0 (0) — keloid formation at sternum

LIMITATIONS AND CAVEATS:
This is a small study and a multi-center study is recommended. In spite of randomization the BoneSeal®, group was younger than the Ostene® group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT03085017/Prot_SAP_001.pdf